CLINICAL TRIAL: NCT03229668
Title: Effect of Pregabalin Administration on Catheter- Related Bladder Discomfort in Urological Surgical Operations
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saint Savvas Anticancer Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgia Micha, Anesthesiologist,MD, MSc, PhD, Saint Savvas Anticancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRBD urologic operations
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pregabalin on Catheter Related Bladder Discomfort
Keywords: urinary bladder; urinary catheters; pregabalin
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind,randomized, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Placebo Comparator): Administration of a placebo capsule 1 hour prior to the surgical operation
  Interventions: Drug: Placebo oral capsule
- Group II (Experimental): Administration of 75mg of pregabalin 1 hour prior to the surgical operation
  Interventions: Drug: Pregabalin Oral Capsule [Lyrica] 75mg
- Group III (Experimental): Administration of 150mg of pregabalin 1 hour prior to the surgical operation
  Interventions: Drug: Pregabalin Oral Capsule [Lyrica] 150 mg

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo oral capsule administered 1 hour prior to the surgical operation
  Arms: Group I
Drug: Pregabalin Oral Capsule [Lyrica] 75mg — Pregabalin Oral Capsule [Lyrica] 75 mg administered 1 hour prior to the surgical operation
  Other Names: Pregabalin
  Arms: Group II
Drug: Pregabalin Oral Capsule [Lyrica] 150 mg — Pregabalin Oral Capsule [Lyrica] 150 mg administered 1 hour prior to the surgical operation
  Other Names: Pregabalin
  Arms: Group III

SUMMARY:
The aim of this study is to assess the effect of pregabalin administration on catheter-related bladder discomfort (CRBD). The study group includes patients that are about to be subjected to urological operations because of the high incidence of CRBD observed in this kind of surgical population.

ELIGIBILITY:
Inclusion Criteria:

* All patients about to be subjected to urinary operations
* Signed informed consent

Exclusion Criteria:

* Preoperative urinary bladder/kidney dysfunction as a result of spinal cord pathology
* History of overactive ((urinary frequency>3 times at night and >8 times in 24 hours), neurogenic bladder
* End stage renal failure
* Central nervous system dysfunction
* Mental illness/ substance abuse
* Sensitivity to pregabalin
* Preoperative administration of pregabalin for other indications
* Recent bladder catheterization <3 months

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Percentage of postsurgical catheter-related bladder discomfort after preoperative pregabalin administration | Change from preoperative status to postoperative one at 0, 1, 2, 6, 24 hours postoperatively
  Assessment of discomfort will be made by a scale of four (1=no discomfort, 2=mild discomfort reported on questioning only, 3=moderate discomfort, urge to pass urine reported by the patient without questioning, 4= severe discomfort, urge to pass urine accompanied by behavioral responses, such as flailing limbs, strong vocal responses or attempts to pull the catheter out)

SECONDARY OUTCOMES:
Postoperative pain assessed by NPRS scale (Numeric Pain Rating Scale) | Total amount of analgesics in morphine analogues administered in the first 24 hours postoperatively
  The goal is to achieve pain scores<3 as these are assessed by the NPRS scale. In order to achieve that we will record the total amount of milligrams of analogues of morphine administered in the first 24 hours postoperatively
Adverse effects of the drug | All adverse effects observed in the first 24 hours postoperatively
  Postoperative nausea and vomiting, confusion, vertigo, blurred vision, dry mouth,sedation, dizziness
Assessment of postoperative sedation | In the operating theatre immediately after patient's extubation
  The Ramsay Sedation Scale is used to measure different levels of sedation in medical patients (1=Patient is anxious and agitated or restless, or both 2=Patient is co-operative, oriented, and tranquil, 3=Patient responds to commands only, 4=Patient exhibits brisk response to light glabellar tap or loud auditory stimulus, 5=Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus, 6=Patient exhibits no response)

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, Prof Of Anesthesiology, Study Chair — University of Thessaly, Medical School, Anesthesiology Clinic
Locations (2):
- Greece (2):
  - Anticancer Hospital of Athens "Saint Savvas", Athens
  - University of Thessaly, Medical School, Volos

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agarwal A, Dhiraaj S, Singhal V, Kapoor R, Tandon M. Comparison of efficacy of oxybutynin and tolterodine for prevention of catheter related bladder discomfort: a prospective, randomized, placebo-controlled, double-blind study. Br J Anaesth. 2006 Mar;96(3):377-80. doi: 10.1093/bja/ael003. Epub 2006 Jan 16. PMID 16415311
- [Background] Srivastava VK, Agrawal S, Kadiyala VN, Ahmed M, Sharma S, Kumar R. The efficacy of pregabalin for prevention of catheter-related bladder discomfort: a prospective, randomized, placebo-controlled double-blind study. J Anesth. 2015 Apr;29(2):212-6. doi: 10.1007/s00540-014-1911-x. Epub 2014 Sep 9. PMID 25200037
- [Background] Tauzin-Fin P, Stecken L, Sztark F. [Catheter-related bladder discomfort in post-anaesthesia care unit]. Ann Fr Anesth Reanim. 2012 Jul-Aug;31(7-8):605-8. doi: 10.1016/j.annfar.2012.03.009. Epub 2012 Jun 29. French. PMID 22749555
- [Background] Bai Y, Wang X, Li X, Pu C, Yuan H, Tang Y, Li J, Wei Q, Han P. Management of Catheter-Related Bladder Discomfort in Patients Who Underwent Elective Surgery. J Endourol. 2015 Jun;29(6):640-9. doi: 10.1089/end.2014.0670. Epub 2014 Dec 9. PMID 25335575
- [Background] Ryu JH, Hwang JW, Lee JW, Seo JH, Park HP, Oh AY, Jeon YT, Do SH. Efficacy of butylscopolamine for the treatment of catheter-related bladder discomfort: a prospective, randomized, placebo-controlled, double-blind study. Br J Anaesth. 2013 Dec;111(6):932-7. doi: 10.1093/bja/aet249. Epub 2013 Jul 17. PMID 23869107
- [Background] Agarwal A, Gupta D, Kumar M, Dhiraaj S, Tandon M, Singh PK. Ketamine for treatment of catheter related bladder discomfort: a prospective, randomized, placebo controlled and double blind study. Br J Anaesth. 2006 May;96(5):587-9. doi: 10.1093/bja/ael048. Epub 2006 Mar 10. PMID 16531445
- [Background] Agarwal A, Yadav G, Gupta D, Singh PK, Singh U. Evaluation of intra-operative tramadol for prevention of catheter-related bladder discomfort: a prospective, randomized, double-blind study. Br J Anaesth. 2008 Oct;101(4):506-10. doi: 10.1093/bja/aen217. Epub 2008 Jul 24. PMID 18653496
- [Background] Nam K, Seo JH, Ryu JH, Oh AY, Lee T, Park HP, Jeon YT, Hwang JW. Randomized, clinical trial on the preventive effects of butylscopolamine on early postoperative catheter-related bladder discomfort. Surgery. 2015 Feb;157(2):396-401. doi: 10.1016/j.surg.2014.05.017. Epub 2014 Oct 8. PMID 25304838